CLINICAL TRIAL: NCT06676696
Title: A Multi-centre, Open, Prospective, Randomized, Parallel-group, 24-month Study to Compare the Outcome of Receiving Continued Immunosuppression Versus Stopping Immunosuppression at 6 Months to Safely Prevent Human Leukocyte Antigen (HLA) Sensitization in Patients With Late Renal Graft Failure
Brief Title: Study to Compare the Outcome of Receiving Continued Immunosuppression Versus Stopping Immunosuppression at 6 Months to Safely Prevent Human Leukocyte Antigen (HLA) Sensitization in Patients With Late Renal Graft Failure
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREVSENSI; 2023-506879-98-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Renal Failure , Chronic; Graft Failure; Graft Rejection; Allograft; Renal Failure Chronic Requiring Dialysis
Keywords: Renal failure; immunosuppressor; HLA sensitization; Graft failure; Calcineurin inhibitors
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency | interventions — Calcineurin Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (Active Comparator)
  Interventions: Drug: Calcineurin inhibitor withdrawal at 6 months
- Investigational arm (Active Comparator)
  Interventions: Drug: Continue low dose calcineurin inhibitor (CNI)

INTERVENTIONS:
Drug: Continue low dose calcineurin inhibitor (CNI) — CNI dose (tacrolimus or cyclosporine) will be adjusted to maintain low tacrolimus or cyclosporine whole blood trough levels from month 3 to month 24 or End of Study
  Arms: Investigational arm
Drug: Calcineurin inhibitor withdrawal at 6 months — CNI dose (tacrolimus or cyclosporine) will be reduced to one-half on month 3 visit and completely withdrawn on month 6 visit.
  Arms: Control Arm

SUMMARY:
The goal of this clinical trial is to compare the degree of HLA sensitization at 2 years in patients with late renal graft failure (> 3 months) when receiving reduced immunosuppressant treatment versus stopping immunosuppression at 6 months.

The main question this study aims to answer is:

Does maintaining long-term immunosuppression in patients with a late renal graft failure (> 3 months) safely reduce the risk of HLA sensitization?

To answer this question, patients will be assigned to a control arm or investigational arm:

* Patients assigned to the control arm will receive standard treatment, in which immunosuppressant treatment is withdrawn after 6 months.
* Patients assigned to the investigatonal arm will continue immunosuppressant treatment at low doses for 2 years.

Patients recruited in this clinical trial will be followed for up to 2 years. During this time, patients will visit the clinic every 3 months for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be able to understand and provide written informed consent
* Patients older than 18 years who had received at least one previous renal transplant
* Patients with a retained kidney graft failed for any reason which survived at least 3 months
* Patients on dialysis, either hemodialysis or peritoneal dialysis. Patients can be on dialysis for a maximum of 6 months at the time of randomization, as long as the patients have taken an uninterrupted immunosuppressive regimen of calcineurin inhibitors (tacrolimus or cyclosporine) and steroids since dialysis was restarted
* Patients already relisted or candidates to relist to deceased donor kidney transplantation according to the treating physician criteria
* Patients taking immunosuppressants tacrolimus or cyclosporine
* cPRA at the time of randomization ≤ 90%

Exclusion Criteria:

* Patients who have received another solid organ transplantation (liver, lung, heart or pancreas)
* Patients waiting for a living related / unrelated kidney transplant
* Graft survival of the failed graft lower than 3 months
* Patients in dialysis more than 6 months at the time of randomization
* Patients not accomplishing criteria to relist in the transplantation list according to the treating physician criteria
* Pregnant women
* Females of childbearing age who have not used or do not plan to use acceptable birth control measures, for the duration of the study. Patients should use one of the acceptable birth control measures recommended in the document "Recommendations related to contraception and pregnancy testing in clinical trials" published by the Clinical Trials Facilitation and Coordination Group (CTFG) (version 1.1, published 21/09/2020). Recommended birth control measures include oral, injected or implanted hormonal contraceptive, barrier methods (condom or diaphragm with spermicide), intrauterine device, surgical sterilization, transdermal delivery, or sexual abstinence. If sexually active, the subject must have been using one of the accepted birth control methods at least one month prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Degree of HLA sensitization | 2 years
  The difference between the two treatment arms in the degree of HLA sensitization at 2-years measured as cPRA (%).

SECONDARY OUTCOMES:
Mortality for any reason | 2 years
  The difference between the two treatment arms at 2-years on mortality for any reason
Days of hospitalization for any reason | 2 years
  The difference between the two treatment arms at 2-years on days of hospitalization for any reason
Percentage of patients effectively relisted during follow-up | 2 years
  The difference between the two treatment arms at 2-years on percentage of patients effectively relisted during follow-up
Percentage of patients transplanted | 2 years
  The difference between the two treatment arms at 2-years on percentage of patients transplanted
Percentage of patients delisted for any reason | 2 years
  The difference between the two treatment arms at 2-years on percentage of patients delisted for any reason
Incidence of infection | 2 years
  The difference between the two treatment arms at 2-years on incidence of infection
Incidence of cardiovascular events | 2 years
  The difference between the two treatment arms at 2-years on incidence of cardiovascular events
Incidence of cancer | 2 years
  The difference between the two treatment arms at 2-years on incidence of cancer
Incidence of graft-intolerance syndrome requiring graft nephrectomy or percutaneous embolization of the non-functioning graft | 2 years
  The difference between the two treatment arms at 2-years incidence of graft-intolerance syndrome requiring graft nephrectomy or percutaneous embolization of the non-functioning graft
Erythropoietin resistance index | 2 years
  The difference between the two treatment arms at 2-years on erythropoietin resistance index
Residual renal function | 2 years
  The difference between the two treatment arms at 2-years on residual renal function
Number of circulating memory B-cells | 2 years
  The difference between the two treatment arms at 2-years on number of circulating memory B-cells
Adverse events | 2 years
  The difference in the incidence of adverse events (AE) in the two treatment arms

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Vall D'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided